CLINICAL TRIAL: NCT00022672
Title: A Randomized, Open-label Study of the Effect of Herceptin Plus Arimidex Compared With Arimidex Alone on Progression-free Survival in Patients With HER2-positive and Hormone-receptor Positive Metastatic Breast Cancer
Brief Title: A Study to Evaluate the Efficacy and Safety of Herceptin® (Trastuzumab) in Combination With Arimidex® (Anastrozole) an Aromatase Inhibitor Compared to Arimidex® Alone in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO16216; NCT00112450 (obsolete NCT alias)
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Results first posted 2013-06-13 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Anastrozole

ARMS (2):
- trastuzumab + anastrozole (Experimental): Trastuzumab 4 mg/kg loading dose intravenous (iv) over 90 minutes, followed by weekly doses of 2 mg/kg iv over 30 minutes plus 1 mg oral dose of anastrozole every day for 24 Months in the Main phase and in the Extension Phase.
  Interventions: Drug: trastuzumab (Herceptin®); Drug: anastrazole (Arimidex®)
- anastrozole (Active Comparator): 1 mg oral dose of anastrozole every day for 24 Months in the Main phase. In the Extension Phase participants could cross-over to also receive trastuzumab 4 mg/kg initial loading dose intravenous (iv) over 90 minutes, followed by weekly doses of 2 mg/kg iv over 30 minutes.
  Interventions: Drug: anastrazole (Arimidex®)

INTERVENTIONS:
Drug: trastuzumab (Herceptin®) — 4mg/kg iv loading dose, followed by 2mg/kg iv weekly
  Other Names: Herceptin®
  Arms: trastuzumab + anastrozole
Drug: anastrazole (Arimidex®) — 1 mg tablet taken orally daily
  Other Names: Arimidex®

SUMMARY:
This 2 arm study assessed the safety and efficacy of adding intravenous trastuzumab (Herceptin®) to daily oral anastrozole (Arimidex®) tablets as first- and second-line treatment in postmenopausal patients with human epidermal growth factor receptor-2 (HER2) overexpressing metastatic breast cancer (ER+ve and/or PR+ve). Patients were randomized to receive either anastrazole 1 mg per os (po) daily, or anastrazole 1 mg po daily + a loading dose of Herceptin® 4 mg/kg intravenous (iv) followed by weekly doses of Herceptin® 2 mg/kg iv. The anticipated time on study treatment was until disease progression, and the target sample size was 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women;
* metastatic breast cancer suitable for endocrine therapy;
* positive hormone receptor status;
* Human epidermal growth factor receptor 2 (HER2) overexpression.

Exclusion Criteria:

* patients on hormone replacement therapy;
* previous chemotherapy for metastatic disease;
* uncontrolled cardiac disease and history of cardiac failure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2001-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (112):
- United States (19):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Los Angeles, California
  - Vallejo, California
  - Gainsville, Florida
  - Miami, Florida
  - Plantation, Florida
  - Chicago, Illinois
  - Kansas City, Kansas
  - Scarborough, Maine
  - Detroit, Michigan
  - Omaha, Nebraska
  - Hackensack, New Jersey
  - Albuquerque, New Mexico
  - Santa Fe, New Mexico
  - Rochester, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Hershey, Pennsylvania
- Australia (3):
  - Box Hill
  - Darlinghurst
  - Waratah
- Porto Alegre, Brazil
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Stara Zagora
- Canada (8):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Oshawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- China (3):
  - Beijing
  - Shanghai
  - Wuhan
- France (2):
  - Avignon
  - Nice
- Germany (4):
  - Frankfurt
  - Kiel
  - München
  - Trier
- Hong Kong, Hong Kong
- Budapest, Hungary
- India (7):
  - Ahmedabad
  - Bangalore
  - Chennai
  - Cuttack
  - Ludhiana
  - Mumbai
  - New Delhi
- Israel (5):
  - Haifa
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Tel Aviv
- Genova, Italy
- Vilnius, Lithuania
- Mexico (2):
  - Guadalajara
  - Mexico City
- Netherlands (2):
  - Amsterdam
  - Rotterdam
- Trondheim, Norway
- Poland (7):
  - Bialystok
  - Bydgoszcz
  - Gliwice
  - Krakow
  - Lodz
  - Szczecin
  - Warsaw
- Russia (7):
  - Barnaul
  - Izhevsk
  - Kazan'
  - Krasnodar
  - Moscow
  - Saint Petersburg
  - Ufa
- South Africa (2):
  - Floracliffe
  - Pretoria
- Spain (7):
  - Barcelona
  - Córdoba
  - Girona
  - Madrid
  - Mataró
  - Reus
  - Valencia
- Sweden (4):
  - Borås
  - Gaelve
  - Örebro
  - Stockholm
- Taiwan (2):
  - Taipei
  - Taoyuan District
- Turkey (Türkiye) (4):
  - Ankara
  - Istanbul
  - Izmir
  - Shhiye, Ankara
- Ukraine (5):
  - Kiev
  - Lviv
  - Odesa
  - Sumy
  - Zaporizhzhya
- United Kingdom (10):
  - Cardiff
  - Edinburgh
  - Guildford
  - Ipswich
  - London
  - Manchester
  - Merseyside
  - Newcastle upon Tyne
  - Southampton
  - Swansea

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 208 participants were randomized. 1 participant did not receive study drug. After the completion of the 24 month Main Phase or disease progression, participants in the anastrozole-alone treatment arm entered the Extension Phase where they received trastuzumab + anastrozole.
Period: Main Phase: 24 Months
Arm/Group | Trastuzumab + Anastrozole | Anastrozole
Started | 103 | 104
Safety Set: Received Study Drug | 103 | 104
Completed | 16 | 4
Not Completed | 87 | 100
Not completed — Adverse Event | 6 | 0
Not completed — Death | 0 | 3
Not completed — Insufficient Therapeutic Response | 75 | 91
Not completed — Violation of Selection Criteria at Entry | 0 | 1
Not completed — Other Protocol Violation | 1 | 0
Not completed — Refused Treatment | 3 | 4
Not completed — Failure to Return | 1 | 1
Not completed — Other | 1 | 0
Period: Extension Phase
Arm/Group | Trastuzumab + Anastrozole | Anastrozole
Started | 14 (2 patients completed Main Phase; but did not enter Extension (1-did not cooperate and 1-withdrew).) | 58
Safety Set: Received Study Drug | 14 | 58
Completed | 11 | 7
Not Completed | 3 | 51
Not completed — Adverse Event | 1 | 3
Not completed — Death | 0 | 1
Not completed — Insufficient Therapeutic Response | 1 | 44
Not completed — Refused Treatment | 0 | 2
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab + Anastrozole | Anastrozole | Total
Number analyzed (Participants) | 103 | 104 | 207
Age Continuous [Mean (Standard Deviation); unit: years] | 57.4 (10.6) | 55.5 (10.7) | 56.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 104 | 207
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was assessed by the investigator based on World Health Organization (WHO) criteria using radiographic tumor evaluations. Disease progression was defined as the appearance of any new lesion not previously identified or an estimated increase of 25% or more in existent bidimensionally or unidimensionally measurable lesions or progression of an existing non-measurable lesion. For bidimensionally measurable malignant lesions with an area of at least 2.0 centimeters squared (cm^2) an increase of 1.0 cm^2 was required and for unidimensionally measurable lesions of 1.0 cm or less an increase of 0.5 cm was required. PFS was defined as the number of days between date of randomization and date of documented disease progression or date of death. Kaplan Meier estimates of PFS are presented.
Time Frame: 24 Months, End of Study (Up to 5 years)
Population: Full analysis population included all randomized participants who received study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab + Anastrozole | Anastrozole
Number analyzed (Participants) | 103 | 104
Months
  24 Months | 4.8 [3.7 to 7] | 2.4 [2 to 4.6]
  End of Study | 5.8 [4.6 to 8.3] | 2.9 [2.1 to 4.5]

2. Secondary Outcome: Percentage of Participants With Clinical Benefit
Description: Clinical Benefit was defined as stable disease for ≥ six months or complete response or partial response.
Time Frame: 24 Months, End of Study (Up to 5 years)
Measure: Number; unit: Percentage of participants
Arm/Group | Trastuzumab + Anastrozole | Anastrozole
Number analyzed (Participants) | 103 | 104
Percentage of participants
  24 Months | 42.7 | 27.9
  End of Study | 45.6 | 30.8

3. Secondary Outcome: Duration of Response at 24 Months
Description: Duration of response was defined as the number of days from the day complete response or partial response was first noted to the day of progression of disease, death or last follow-up.
Time Frame: 24 Months
Population: Participants from the Full Analysis population (all randomized participants who received study drug) evaluable for response.
Measure: Median (Full Range); unit: Months
Arm/Group | Trastuzumab + Anastrozole | Anastrozole
Number analyzed (Participants) | 74 | 73
Months | 9.5 [3.8 to 50.6] | 10.0 [5.3 to 33.1]

4. Secondary Outcome: Time to Response at 24 Months
Description: Time to response was defined as the number of days from the day of randomization to the day complete response or partial response was first noted.
Time Frame: 24 Months
Population: as for outcome 3
Measure: Median (Full Range); unit: Months
Arm/Group | Trastuzumab + Anastrozole | Anastrozole
Number analyzed (Participants) | 74 | 73
Months | 2.0 [1.4 to 12.1] | 2.0 [1.7 to 4.1]

5. Secondary Outcome: Overall Survival at 24 Months
Description: Overall Survival is defined as the number of days from randomization to death.
Time Frame: 24 Months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab + Anastrozole | Anastrozole
Number analyzed (Participants) | 103 | 104
Months | 28.5 [22.8 to 42.4] | 23.9 [18.2 to 37.4]

6. Secondary Outcome: Percentage of Participants With Two-Year Survival
Time Frame: 24 Months
Population: Full Analysis Population included all randomized participants who received study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Trastuzumab + Anastrozole | Anastrozole
Number analyzed (Participants) | 103 | 104
Percentage of participants | 52.4 | 45.2

7. Secondary Outcome: Percentage of Participants With Overall Tumor Response at 24 Months
Description: Tumor Response levels were determined by the investigator and an Independent Response Evaluation Committee and Reconciled. Overall Response was defined as either complete response or partial response.
Time Frame: 24 Months
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Trastuzumab + Anastrozole | Anastrozole
Number analyzed (Participants) | 74 | 73
Percentage of participants | 20.3 | 6.8

8. Secondary Outcome: Percentage of Participants With Best Tumor Response at 24 Months
Description: Tumor Response levels were determined by the investigator and an Independent Response Evaluation Committee and Reconciled. Best Response was defined as the best response a patient achieves in the study.
Time Frame: 24 Months
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Trastuzumab + Anastrozole | Anastrozole
Number analyzed (Participants) | 74 | 73
Percentage of participants
  Complete Response | 0.0 | 0.0
  Partial Response | 20.3 | 6.8
  Stable Disease | 37.8 | 38.4
  Progressive Disease | 40.5 | 49.3
  Response not assessed | 1.4 | 5.5

9. Secondary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status at Final Visit Compared to Baseline
Description: Participants rated their performance status using the ECOG Questionnaire on the following scale: 0=Fully active, perform all pre-disease activities without restriction; 1=Restricted in physically strenuous activity but ambulatory, carry out work of a light or sedentary nature; 2=Ambulatory, capable of self-care, unable to carry out any work activities, up and about more than >50% of waking hours; 3=Capable of limited self-care, confined to bed or chair >50% of waking hours; 4=Completely disabled, not capable of any self-care, totally confined to bed or chair; 5=Dead.
  The percentage of participants in the following categories:
  Improved: Score decrease from baseline. Unchanged: Score the same as baseline. Worse: Score increase from baseline.
Time Frame: Baseline, Final Visit (Up to 24 Months)
Population: Participants from the Full Analysis Population (includes all randomized participants who received study drug) with data available for analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | Trastuzumab + Anastrozole | Anastrozole
Number analyzed (Participants) | 68 | 73
Percentage of participants
  Improved | 10.3 | 4.1
  No Change | 67.6 | 64.4
  Worse | 22.1 | 31.5

10. Secondary Outcome: Duration of Response at End of Study
Description: as for outcome 3
Time Frame: End of Study (Up to 5 years)
Population: as for outcome 3
Measure: Median (Full Range); unit: Months
Arm/Group | Trastuzumab + Anastrozole | Anastrozole
Number analyzed (Participants) | 103 | 104
Months | 12.3 [3 to 59.1] | 8.2 [2.6 to 60.5]

11. Secondary Outcome: Time to Response at End of Study
Description: as for outcome 4
Time Frame: End of Study (Up to 5 years)
Population: as for outcome 3
Measure: Median (Full Range); unit: Months
Arm/Group | Trastuzumab + Anastrozole | Anastrozole
Number analyzed (Participants) | 103 | 104
Months | 2.4 [1.7 to 12.1] | 2.1 [1.3 to 5.1]

12. Secondary Outcome: Percentage of Participants With Overall Tumor Response at End of Study
Description: as for outcome 7
Time Frame: End of Study (Up to 5 years)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Trastuzumab + Anastrozole | Anastrozole
Number analyzed (Participants) | 103 | 104
Percentage of participants | 22.3 | 8.7

13. Secondary Outcome: Percentage of Participants With Best Tumor Response at End of Study
Description: as for outcome 8
Time Frame: End of Study (Up to 5 years)
Population: Full Analysis Population includes all randomized participants who received study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Trastuzumab + Anastrozole | Anastrozole
Number analyzed (Participants) | 103 | 104
Percentage of participants
  Complete Response | 1.0 | 3.8
  Partial Response | 21.4 | 4.8
  Stable Disease | 47.6 | 40.4
  Progressive Disease | 28.1 | 46.2
  Response not assessed | 1.9 | 4.8

14. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with adverse events as a measure for safety as assessed by the collection of adverse events, laboratory tests for Hematology and Serum Chemistry, clinical assessments and cardiac monitoring.
Time Frame: Throughout the Study (Up to 5 years)
Population: Safety population included all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Trastuzumab + Anastrozole | Anastrozole
Number analyzed (Participants) | 103 | 104
Participants | 90 | 68

ADVERSE EVENTS:
Groups:
- Anastrozole: 1 mg oral dose of anastrozole every day for 24 Months in the Main phase.
- Anastrozole (After Start of Trastuzumab): 1 mg oral dose of anastrozole every day for 24 Months in the Main phase. In the Extension Phase participants could cross-over to also receive trastuzumab 4 mg/kg initial loading dose intravenous (iv) over 90 minutes, followed by weekly doses of 2 mg/kg iv over 30 minutes.
Arm/Group | Trastuzumab + Anastrozole | Anastrozole | Anastrozole (After Start of Trastuzumab)
Serious Adverse Events (participants affected / at risk) | 25/103 | 6/104 | 8/58
Other Adverse Events (participants affected / at risk) | 89/103 | 68/104 | 40/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + Anastrozole (N=103) | Anastrozole (N=104) | Anastrozole (After Start of Trastuzumab) (N=58)
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Malaria (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0 | 0
Chest pain (General disorders) | 3 | 0 | 0
Pain (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
Venous insufficiency (Vascular disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + Anastrozole (N=103) | Anastrozole (N=104) | Anastrozole (After Start of Trastuzumab) (N=58)
Constipation (Gastrointestinal disorders) | 11 | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 20 | 8 | 8
Nausea (Gastrointestinal disorders) | 15 | 5 | 5
Vomiting (Gastrointestinal disorders) | 21 | 5 | 5
Chills (General disorders) | 15 | 0 | 3
Fatigue (General disorders) | 22 | 10 | 4
Oedema peripheral (General disorders) | 7 | 2 | 4
Pyrexia (General disorders) | 17 | 6 | 4
Influenza (Infections and infestations) | 7 | 4 | 1
Nasopharyngitis (Infections and infestations) | 17 | 2 | 2
Weight decreased (Investigations) | 9 | 4 | 3
Weight increased (Investigations) | 9 | 4 | 1
Anorexia (Metabolism and nutrition disorders) | 7 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 9 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 7 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 11 | 6 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 4 | 3
Dizziness (Nervous system disorders) | 10 | 4 | 2
Headache (Nervous system disorders) | 14 | 6 | 2
Depression (Psychiatric disorders) | 6 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 6 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 9 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 2 | 6
Rash (Skin and subcutaneous tissue disorders) | 6 | 6 | 1
Hot flush (Vascular disorders) | 9 | 3 | 0
Hypertension (Vascular disorders) | 6 | 4 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 3
Lacrimation increased (Eye disorders) | 1 | 0 | 4
Mucosal inflammation (General disorders) | 5 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.